CLINICAL TRIAL: NCT06448832
Title: Relationship of Muscular Agenesis: Thin Plantar and Palmar Long as a Biomarker of Injury and Performance Marker in the Lower Limb and Upper Limb Respectively
Acronym: MA-TP-PL
Status: Not yet recruiting | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, JJ JIMENEZ-REJANO, PhD, University of Seville
Other Study IDs: Muscular Agenesis Thin plantar
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Abnormality, Congenital
Keywords: muscle agenesis; thin plantar; force; injuries; musculoskeletal palmar long; performance
MeSH Terms: conditions — Congenital Abnormalities; Wounds and Injuries | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Agenesis Group: Subjects with the presence of muscular agenesis of the plantar muscle and palmaris longus.
  Interventions: Diagnostic Test: Ultrasound
- Non-agenesis Group: Subjects without the presence of muscular agenesis of the plantar muscle and palmaris longus.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — An ultrasound examination of the musculature of the plantar muscle and long palmar muscle is performed to determine their presence or absence.

SUMMARY:
This study investigates muscle agenesis, specifically the absence of the palmaris longus and plantaris muscles, and its effects on injury risk, strength, and performance. Muscle injuries are common in sports, and the presence or absence of certain muscles can impact biomechanics and injury susceptibility. The study involves 132 subjects, divided into those with and without muscle agenesis, assessing injuries with the Nordic and CMDQ questionnaires and measuring strength with dynamometers. Results aim to clarify the controversial impact of muscle agenesis on functional disability and performance adaptation in the scientific literature.

DETAILED DESCRIPTION:
Background. This study examines muscle agenesis, a congenital condition that involves the absence of a muscle, focusing on the palmaris longus and plantaris muscles. The prevalence of palmaris longus agenesis varies significantly, and there is debate about whether its absence results in functional disability or is a predictor of injuries. Muscle injuries account for one-third of sports injuries and more than 30% of all musculoskeletal system injuries. The presence or absence of certain muscles can influence the body's biomechanics and, therefore, susceptibility to injuries, as muscles play a crucial role in generating force and coordination, hence movement. The absence of certain muscles may require other muscles to compensate, which could affect the efficiency and performance capacity in certain body areas. However, in many cases, the absence of a muscle may not have a significant effect on performance, as other muscles can adapt to perform its function. This study seeks to provide clarity in this area of research due to the existing controversy in the scientific literature.

Objectives. To determine if muscle agenesis influences the development of injuries and its impact on strength and performance.

Material and methods. An observational analytical cross-sectional study was conducted with 132 subjects divided into one group of 66 subjects with muscle agenesis and another group of 66 subjects without muscle agenesis. The primary variable is the presence of upper and lower limb injuries measured using the Nordic and CMDQ questionnaires, and the secondary variable is upper limb strength measured with a dynamometer in palmar flexion and hand grip tests; and lower limb strength measured with a dynamometer in plantar flexion and vertical jump tests. The measurements were taken over 1 hour and 30 minutes during two days, with a 48-hour interval between the measurements of the upper and lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who lead a sedentary lifestyle or who are not used to doing physical training on a regular basis (more than 2 h/week).
* People between 18 and 80 years old.

Exclusion Criteria:

* Individuals with an ongoing oncological process.
* People with an active infectious process.
* Subjects with psychiatric disorders.
* Individuals with intellectual disorders that prevent understanding of the intervention.
* People with judicial incapacity.
* Patients diagnosed with fibromyalgia.
* Pregnancy or probability of pregnancy.
* Individuals with sensory impairments in the hand that prevent manual pressure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with and without muscle agenesis.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Presence of injury | At the start of the study (at baseline, 0 week).
  Presence of injury related to the upper and lower limb.

SECONDARY OUTCOMES:
Strength | At the start of the study (at baseline, 0 week)
  Upper and lower limb strength

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Garcia-Luna, MSc, Principal Investigator — University of Alcala; Jose-Jesus Jimenez-Rejano, PhD, Principal Investigator — University of Seville
Locations (1):
- Campus Científico-Tecnológico UAH. Av. de León, 3A, Alcalá de Henares, Madrid, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balsalobre-Fernandez C, Glaister M, Lockey RA. The validity and reliability of an iPhone app for measuring vertical jump performance. J Sports Sci. 2015;33(15):1574-9. doi: 10.1080/02640414.2014.996184. Epub 2015 Jan 2. PMID 25555023
- [Background] Ioannis D, Anastasios K, Konstantinos N, Lazaros K, Georgios N. Palmaris Longus Muscle's Prevalence in Different Nations and Interesting Anatomical Variations: Review of the Literature. J Clin Med Res. 2015 Nov;7(11):825-30. doi: 10.14740/jocmr2243w. Epub 2015 Sep 25. PMID 26491493
- [Background] Vanhoenacker FM, Desimpel J, Mespreuve M, Tagliafico A. Accessory Muscles of the Extremities. Semin Musculoskelet Radiol. 2018 Jul;22(3):275-285. doi: 10.1055/s-0038-1641575. Epub 2018 May 23. PMID 29791956
- [Background] Martinoli C, Perez MM, Padua L, Valle M, Capaccio E, Altafini L, Michaud J, Tagliafico A. Muscle variants of the upper and lower limb (with anatomical correlation). Semin Musculoskelet Radiol. 2010 Jun;14(2):106-21. doi: 10.1055/s-0030-1253155. Epub 2010 May 18. PMID 20486022
- [Background] Eric M, Koprivcic I, Vucinic N, Radic R, Krivokuca D, Leksan I, Selthofer R. Prevalence of the palmaris longus in relation to the hand dominance. Surg Radiol Anat. 2011 Aug;33(6):481-4. doi: 10.1007/s00276-010-0751-0. Epub 2010 Nov 24. PMID 21107568
- [Background] Dabrowski K, Stankiewicz-Jozwicka H, Kowalczyk A, Markuszewski M, Ciszek B. Musculus Palmaris Longus: Influence on Playing Capability of Keyboard Musicians - Preliminary Report. Front Psychol. 2018 Aug 13;9:1460. doi: 10.3389/fpsyg.2018.01460. eCollection 2018. PMID 30150961
- [Background] Vucinic N, Eric M, Savic M. How often absence of palmaris longus and functional deficiencyof flexor digitorum superficialis occurs ? Acta Orthop Belg. 2016 Aug;82(2):405-411. PMID 27682306
- [Background] Amaral JF, Mancini M, Novo Junior JM. Comparison of three hand dynamometers in relation to the accuracy and precision of the measurements. Rev Bras Fisioter. 2012 Jun;16(3):216-24. doi: 10.1590/s1413-35552012000300007. PMID 22801514
- [Background] Chamorro C, Armijo-Olivo S, De la Fuente C, Fuentes J, Javier Chirosa L. Absolute Reliability and Concurrent Validity of Hand Held Dynamometry and Isokinetic Dynamometry in the Hip, Knee and Ankle Joint: Systematic Review and Meta-analysis. Open Med (Wars). 2017 Oct 17;12:359-375. doi: 10.1515/med-2017-0052. eCollection 2017. PMID 29071305
- [Background] Pua YH, Wrigley TV, Cowan SM, Bennell KL. Intrarater test-retest reliability of hip range of motion and hip muscle strength measurements in persons with hip osteoarthritis. Arch Phys Med Rehabil. 2008 Jun;89(6):1146-54. doi: 10.1016/j.apmr.2007.10.028. PMID 18503813
- [Background] Arnold CM, Warkentin KD, Chilibeck PD, Magnus CR. The reliability and validity of handheld dynamometry for the measurement of lower-extremity muscle strength in older adults. J Strength Cond Res. 2010 Mar;24(3):815-24. doi: 10.1519/JSC.0b013e3181aa36b8. PMID 19661831